CLINICAL TRIAL: NCT06804161
Title: SGLT2 Inhibition for Cardiovascular Endpoint Reduction in Hypertension
Acronym: SGLT2-HYPE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Dr. med. Ingo Eitel (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Ingo Eitel, Head of department of medical clinic II, University of Luebeck
Organization: University of Luebeck (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 724154
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Atrial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGLT2 Arm (Experimental)
  Interventions: Drug: SGLT2
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SGLT2 — 10 mg
  Arms: SGLT2 Arm
Drug: Placebo — 1 tablet
  Arms: Placebo

SUMMARY:
Hypertension (HTN) is a leading cause of cardiovascular disease (CVD). Despite existing therapies, patients with HTN still face substantial risks, due to pre-existing and ongoing end-organ damage due, in part, to inadequate blood pressure (BP) control. SGLT2 inhibitors (SGLT2i) are recommended for both type-2 diabetes and heart failure to reduce morbidity and mortality. SGLT2i reduce BP and might also improve outcomes for HTN by reducing end-organ damage through diverse other actions. However, confirmation that SGLT2i are clinically useful for the management of HTN is required to change guidelines and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60 years
2. Systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg in two measurements on different days for newly diagnosed hypertension, or through one measurement at the screening visit for patients with an existing diagnosis of hypertension.
3. A history of at least one CV event (myocardial infarction* or stroke*; stable angina or clinical evidence of coronary heart disease; peripheral arterial disease; transient ischemic attack)

or

The presence of at least one cardiovascular risk factor (current smoking of more than one cigarette per day during at least 1 year; LDL-cholesterol > 4,0 mmol/l, Age ≥ 75 years, ESC HeartScore > 15%, BMI > 32 kg/m2)

*excluding patients with myocardial infarction or stroke within preceding 3 months

Exclusion Criteria:- Known secondary cause of hypertension

* Myocardial infarction or stroke within the previous 3 months
* Symptomatic heart failure (including HFrEF, HFmEF, HFpEF)
* History of Diabetes mellitus
* History of ketoacidosis
* Hepatic impairment (aspartate transaminase [AST] or alanine transaminase [ALT] >3x the upper limit of normal [ULN])
* eGFR <25 mL/min/1.73 m2 (CKD-EPICr 2021 formula) at Visit 1
* Receiving therapy with an SGLT2i within 8 weeks prior to randomization or previous intolerance to an SGLT2i
* Participation in another clinical study with an investigational product during the last month prior to enrolment
* Known allergy or hypersensitivity to SGLT2i
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Any medical condition - outside the renal and CV disease area - with a life expectancy of less than 2 years based on investigator's clinical judgement
* Active malignancy requiring treatment at the time of visit 1 (with the exception of successfully treated basal cell or treated squamous cell carcinoma)
* Inability to give informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2032-05-30 (Estimated); Study Completion 2032-05-30 (Estimated)

PRIMARY OUTCOMES:
Time until first occurrence of | 7 Years

OTHER OUTCOMES:
Safety endpoints | 7 Years
  * AE (general)
  * AE leading to treatment discontinuation
  * SAE
  * AE of special interest (AESI): including volume depletion, hypotension, metabolic acidosis and ketoacidosis

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Eitel, Prof. Dr., Principal Investigator — Universitätsklinikum Schleswig-Holstein - Campus Lübeck
Locations (1):
- Universität zu Lübeck, Lübeck, Schleswig-Holstein, Germany